CLINICAL TRIAL: NCT04272762
Title: A Randomized Sham-controlled Study of Pulmonary Vein Isolation in Symptomatic Atrial Fibrillation (The SHAM-PVI Study)
Brief Title: A Randomized Sham-controlled Study of Pulmonary Vein Isolation in Symptomatic Atrial Fibrillation
Acronym: SHAM-PVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Sussex Hospitals NHS Trust (Other)
Collaborators: Eastbourne Cardiology Research Charity Fund (Unknown); Medtronic (Industry)
Responsible Party: Principal Investigator, Rick Veasey, Principal Investigator, East Sussex Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 274347
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Ablation; Cryoablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Cryosurgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ablation (Active Comparator): pulmonary vein isolation
  Interventions: Procedure: Cryoablation
- Placebo (Placebo Comparator): placebo procedure
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Cryoablation — Pulmonary vein isolation with cryoablation
  Arms: Ablation
Procedure: Placebo — Placebo procedure
  Arms: Placebo

SUMMARY:
This is a double blinded randomised placebo-controlled trial comparing the effects of catheter ablation (Cryoablation) versus a placebo procedure on atrial fibrillation burden, symptoms and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Symptomatic paroxysmal or persistent atrial fibrillation despite at least one antiarrhythmic drug (AAD Type I or III, β-blocker or AAD intolerance).
* Referred for catheter ablation

Exclusion Criteria:

* Long term persistent AF (continuous episode lasting more than 1)
* Prior left atrium catheter or surgical atrial fibrillation ablation
* Patients with other arrhythmias requiring ablative therapy
* Left atrium (LA) ≥5.5 cm
* Any cardiac surgery or percutaneous coronary intervention (PCI) within three months prior to enrolment.
* Awaiting cardiac surgery or PCI
* Myocardial infarction within three months prior to enrolment.
* Stroke or transient ischemic attack (TIA) within three months prior to enrolment
* Unstable angina
* Any significant congenital heart defect corrected or not (including atrial septal defects or PV abnormalities) but not including patent foramen ovale.
* Any condition contraindicating chronic anticoagulation
* Any untreated or uncontrolled hyperthyroidism or hypothyroidism
* Severe chronic kidney disease (stage V, requiring or almost requiring dialysis, glomerular filtration rate (GFR) < 15 ml / min)
* Patients with metallic prosthetic valves
* Pregnant or breastfeeding women
* Medical conditions limiting expected survival to <1 year
* History of claustrophobia or panic attacks
* Left ventricular ejection fraction (LVEF) less than 35%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation burden using continuous monitoring | 6 months

SECONDARY OUTCOMES:
Time to symptomatic atrial tachyarrhythmia stratified by length of episode | 6 months
Time to asymptomatic atrial tachyarrhythmia stratified by length of episode | 6 months
Number of atrial arrhythmia ( symptomatic and asymptomatic) episodes stratified by length of episode | 6 months
Change in AF specific quality of life score between each group (AF-PROMS) | Baseline and 6 months
Change in health related quality of life in each group (36-Item Short Form Survey Instrument ) | Baseline and 6 months
Comparison of medical treatment ( Antiarrhythmic drug use) | 6 months
Comparison of unscheduled use of health care services | 6 months
Number of procedure related complications / adverse events | 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Mid and South Essex NHS Foundation Trust / The Essex Cardiothoracic Centre, Basildon
  - Eastbourne District General Hospital, Eastbourne
  - Conquest Hospital, Saint Leonards-on-Sea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dulai R, Furniss SS, Sulke N, Freemantle N, Lambiase PD, Farwell D, Srinivasan NT, Tan S, Patel N, Graham A, Veasey RA. A randomized sham-controlled study of pulmonary vein isolation in symptomatic atrial fibrillation (The SHAM-PVI study): Study design and rationale. Clin Cardiol. 2023 Aug;46(8):973-980. doi: 10.1002/clc.24066. Epub 2023 Jun 13. PMID 37309845
- [Derived] Dulai R, Sulke N, Freemantle N, Lambiase PD, Farwell D, Srinivasan NT, Tan S, Patel N, Graham A, Veasey RA. Pulmonary Vein Isolation vs Sham Intervention in Symptomatic Atrial Fibrillation: The SHAM-PVI Randomized Clinical Trial. JAMA. 2024 Sep 2;332(14):1165-73. doi: 10.1001/jama.2024.17921. Online ahead of print. PMID 39221629